CLINICAL TRIAL: NCT00060255
Title: Autologous Blood and Marrow Transplantation for Hematologic Malignancy and Selected Solid Tumors
Brief Title: High-Dose Chemotherapy, Total-Body Irradiation, and Autologous Stem Cell Transplantation or Bone Marrow Transplantation in Treating Patients With Hematologic Cancer or Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000301587; RPCI-DS-9115
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Testicular Germ Cell Tumor; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: stage IV breast cancer; male breast cancer; recurrent malignant testicular germ cell tumor; Waldenstrom macroglobulinemia; childhood acute lymphoblastic leukemia in remission; adult acute lymphoblastic leukemia in remission; recurrent adult acute myeloid leukemia; adult acute myeloid leukemia in remission; recurrent childhood acute myeloid leukemia; childhood acute myeloid leukemia in remission; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent/refractory childhood Hodgkin lymphoma; unspecified adult solid tumor, protocol specific; unspecified childhood solid tumor, protocol specific; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; recurrent breast cancer; primary systemic amyloidosis; refractory multiple myeloma; childhood chronic myelogenous leukemia; atypical chronic myeloid leukemia; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Breast Neoplasms; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Testicular Germ Cell Tumor; Breast Neoplasms, Male; Testicular Neoplasms; Waldenstrom Macroglobulinemia; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Recurrence; Immunoglobulin Light-chain Amyloidosis; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Lymphoma, B-Cell, Marginal Zone; Congenital Abnormalities | interventions — Busulfan; Carboplatin; Carmustine; Cyclophosphamide; Etoposide; Melphalan; Thiotepa; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: busulfan — iv
Drug: carboplatin — iv
Drug: carmustine — iv
Drug: cyclophosphamide — iv
Drug: etoposide — iv
Drug: melphalan — oral
Drug: thiotepa — iv
Procedure: autologous bone marrow transplantation — iv
Procedure: bone marrow ablation with stem cell support — iv
Procedure: peripheral blood stem cell transplantation — iv
Radiation: radiation therapy — body x-ray

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage cancer cells. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with autologous stem cell transplantation or autologous bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: This phase II trial is studying how well eight different high-dose chemotherapy regimens with or without total-body irradiation followed by autologous stem cell transplantation or autologous bone marrow transplantation works in treating patients with hematologic malignancies or solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the morbidity, mortality, and overall outcome in patients with hematologic malignancies, breast cancer, or other chemosensitive solid tumors treated with disease-specific dose-intensive conditioning regimens and autologous peripheral blood or bone marrow transplantation.

OUTLINE: Patients are stratified according to risk group (standard vs high). Standard risk includes acute leukemia in first relapse or second remission; lymphoma in responding first relapse or second remission; or breast cancer at risk for recurrence. High risk includes all others. Patients receive specific conditioning regimens according to diagnosis as outlined below.

Conditioning

* Regimen A (standard risk non-Hodgkin's lymphoma and under 60 years of age)-Etoposide, cyclophosphamide, and total body irradiation (TBI) (VCT): Patients receive etoposide IV continuously over 26 hours beginning on day -5 and cyclophosphamide IV over 2 hours on day -4. Patients undergo TBI on days -3 to -1.
* Regimen B (any risk Hodgkin's lymphoma and under 60 years of age)-Cyclophosphamide, carmustine, and etoposide (CBV): Patients receive etoposide IV continuously over 34 hours beginning on day -8; cyclophosphamide IV over 2 hours on days -7 to -4; and carmustine IV over 2 hours on day -3.
* Regimen C (any risk patient with prior exposure to high-dose etoposide and cyclophosphamide and under 60 years of age)-Melphalan and TBI (MEL/TBI): Patients receive melphalan IV over 30 minutes on day -4. Patients undergo TBI on days -3 to -1.
* Regimen D (multiple myeloma or amyloidosis)-Melphalan only (MEL only): Patients receive melphalan IV over 30 minutes on day -2.
* Regimen E (any patient unable to receive TBI)-Busulfan and cyclophosphamide: Patients receive oral busulfan (or busulfan IV over 2 hours) on days -7 to -4 and cyclophosphamide IV over 2 hours on days -3 and -2.
* Regimen F (any risk breast cancer)-Cyclophosphamide, carboplatin, and thiotepa (STAMP V): Patients receive cyclophosphamide IV over 24 hours, carboplatin IV over 24 hours, and thiotepa IV over 24 hours on days -7 to -4.
* Regimen G (solid tumors other than breast or testicular cancer)-Thiotepa and carboplatin (TT/CARBO): Patients receive thiotepa IV over 2 hours on days -6 and -5 and carboplatin IV continuously over 96 hours beginning on day -6.
* Regimen H (recurrent or primary progressive testicular cancer)-Etoposide and carboplatin (VP/CARBO): Patients receive etoposide IV over 2 hours and carboplatin IV over 30 minutes on days -6 to -4.

Stem Cell Infusion

* In all regimens, patients undergo autologous stem cell infusion on day 0. Treatment continues in the absence of unacceptable toxicity.

PROJECTED ACCRUAL: Approximately 450 patients (50 patients [25 per stratum] per regimen) will be accrued for this study within 10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed hematologic or solid tumor malignancy, including any of the following:

  * Acute myeloid leukemia

    * First remission and not eligible for allogeneic transplantation; recurrent disease after combination chemotherapy with at least 1 standard regimen; or second remission
    * Not eligible for protocol CLB-9620 or CLB-9621
  * Acute lymphoblastic leukemia

    * First complete remission without appropriate allogeneic donor
  * Chronic myelogenous leukemia

    * Chronic, accelerated, or blast phase
  * Lymphoproliferative diseases*

    * Chronic lymphocytic leukemia
    * Multiple myeloma
    * Waldenstrom's macroglobulinemia
    * Low-grade non-Hodgkin's lymphoma (NHL) NOTE: *Recurrent or persistent, symptomatic disease after first-line chemotherapy, or subsequently
  * Amyloidosis

    * Primary or previously treated disease
  * NHL (intermediate- and high-grade)

    * Resistant or recurrent disease after combination chemotherapy with at least 1 standard regimen
    * First remission lymphoblastic or small, non-cleaved cell lymphoma at high risk of relapse

      * CNS disease OR bone marrow disease and lactic dehydrogenase greater than 300 IU/L
  * Hodgkin's lymphoma

    * Resistant or recurrent disease after combination chemotherapy with at least 1 standard regimen
  * Solid tumors

    * High-risk and metastatic breast cancer
    * Testicular cancer that has relapsed OR primary progressive disease that is responding to salvage therapy
    * Other solid tumors that have recurred after conventional therapy OR are at high risk for relapse, and demonstrate chemosensitivity
* Less than 10% marrow tumor present histologically (maximum of 15% involvement allowed if purged)
* Allogeneic marrow transplantation not possible or not desirable for any of the following reasons:

  * Over 60 years of age
  * No compatible donor identified
  * Estimated risk of graft-versus-host disease complications greater than risk of recurrence after autologous bone marrow transplantation
* Patients with disease progression in a site of prior radiotherapy (4,000 cGy or more) are not eligible for total body irradiation (TBI) regimens
* Hormone receptor status:

  * Not specified NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age

* 4 and over (patients 60 years of age and over are not eligible for TBI)

Sex

* Male or female

Menopausal status

* Not specified

Performance status

* Karnofsky 70-100%

Life expectancy

* More than 2 months

Hematopoietic

* WBC greater than 3,000/mm^3*
* Polymorphonuclear leukocyte count greater than 1,500/mm^3*
* Platelet count greater than 75,000/mm^3*
* Marrow cellularity greater than 20%*
* No marrow fibrosis* NOTE: *Before marrow storage

Hepatic

* Bilirubin less than 3 times normal
* Alkaline phosphatase less than 3 times normal
* AST less than 3 times normal
* Hepatitis status known

Renal

* Creatinine clearance at least 50 mL/min (not required for patients with amyloidosis or multiple myeloma)

Cardiovascular

* Ventricular ejection fraction at least 50% by radionuclide ventriculogram or echocardiogram
* No myocardial infarction within the past 6 months
* No congestive heart failure
* No symptomatic angina
* No life-threatening arrhythmia or hypertension

Pulmonary

* DLCO or DLVA at least 50% of predicted (DLCO must be corrected for hemoglobin and/or alveolar ventilation)

Other

* Not pregnant
* HIV negative
* Cytomegalovirus status known
* No active bacterial, viral, or fungal infection
* No active peptic ulcer disease
* No uncontrolled diabetes mellitus
* No serious organ dysfunction unless it is caused by the underlying disease
* No other serious medical or psychiatric illness that would preclude giving informed consent or complying with study requirements

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* See Disease Characteristics
* No prior cumulative nitrosourea dose greater than 600 mg/m^2
* No prior cumulative bleomycin dose greater than 150 units/m^2
* No prior cumulative doxorubicin dose greater than 450 mg/m^2
* No prior cumulative daunorubicin dose greater than 600 mg/m^2
* Patients with prior high-dose cyclophosphamide (greater than 150 mg/kg per cycle) and high-dose etoposide (greater than 2,400 mg/m^2 per cycle) are not eligible for the etoposide/cyclophosphamide/TBI conditioning regimen

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* More than 3 weeks since prior radiotherapy (before blood stem cell harvest)
* Prior cumulative doses of radiotherapy must not exceed the following:

  * Spine/spinal cord: 4,000 cGy
  * Mediastinum: 4,000 cGy
  * Heart: 4,000 cGy
  * Kidney (whole): 1,500 cGy
  * Small bowel: 4,000 cGy
  * Brain: 4,000 cGy
  * Liver (whole): 2,000 cGy
  * Lungs (whole): 1,500 cGy
  * Bone: 5,000 cGy

Surgery

* Not specified

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 1991-12; Primary Completion 2006-08 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Morbidity | +day 100
Mortality | +day 100, +day 360
Overall outcome | every 6 months until death
Response rate | +day 100, +day 360
Toxicity | +day100, +day 360
Disease-free survival | up to 15years
Overall survival | every 6 months until death

CONTACTS AND LOCATIONS:
Overall Officials: Philip L. McCarthy, MD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States